CLINICAL TRIAL: NCT07354906
Title: Prospective Observational Study Evaluating the Efficacy and Safety of Upadacitinib in Giant Cell Arteritis (GCA) With Active Large-vessel Involvement.
Brief Title: Upadacitinib in Giant Cell Arteritis (GCA) With Active Large-vessel Involvement.
Acronym: TILT2
Status: Not yet recruiting | Type: Observational
Sponsor: Groupe français d'étude des Maladies Inflammatoires de loeil (Other)
Responsible Party: Sponsor
Other Study IDs: TILT2; 2025-A02745-44 (Other: ANSM)
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: Giant Cell Arteritis (GCA) .; Upadacitinib; Efficacy
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multicenter cohort evaluating the safety and efficacy of upadacitinib in patients with GCA condition: This is an observational, multicenter cohort evaluating the safety and efficacy of upadacitinib in patients with giant cell arteritis (GCA). Patient treatment and follow-up will be conducted in accordance with routine clinical care. No additional visits or examinations will be added for the purposes of the study. Participants will be followed as part of the usual management of their disease. No modifications will be made (no additional visits, examinations, or questionnaires). The safety and well-being of participants will therefore remain unchanged. Patients will then be followed and managed according to routine care (visits and examinations).
  Routine care includes:
  * A clinical assessment of efficacy and safety at weeks 12, 24, 36, 52, and 104;
  * Oral prednisone treatment at the initial doses recommended by international and French guidelines, in accordance with routine care.

SUMMARY:
Participants will be followed as part of the usual management of their disease. No modifications will be made (no additional visits, examinations, or questionnaires). The safety and well-being of participants will therefore remain unchanged.

The participant will be informed about the study during one of their routine care visits. The information will be provided by the investigator, and the participant's non-opposition to participation in the study will be obtained.

The participant will continue to be followed as part of their usual care.

Data will then be collected from the participant's medical record (including medical reports, original laboratory test results, imaging reports and medical examinations, and nursing records) for the period of participation in the research, solely for the purpose of meeting the objectives of the research.

The data collected will consist of information from the patient's medical record as part of their routine follow-up and will be strictly necessary to address the primary and secondary objectives of the study. The following data will be collected: demographic data (age, sex, weight, height); clinical data (medical history, diagnosed condition, disease activity), treatments, biological data, imaging data, and adverse events. No genetic data will be collected as part of the study. There will be no transfer of data abroad, and no additional questionnaires, examinations, or visits will be added by the research.

DETAILED DESCRIPTION:
This is an observational, multicenter cohort evaluating the safety and efficacy of upadacitinib in patients with giant cell arteritis (GCA). Patient treatment and follow-up will be conducted in accordance with routine clinical care. No additional visits or examinations will be added for the purposes of the study. Participants will be followed as part of the usual management of their disease. No modifications will be made (no additional visits, examinations, or questionnaires). The safety and well-being of participants will therefore remain unchanged.

The participant will be informed about the study during one of their routine care visits. The information will be provided by the investigator, and the participant's non-opposition to participation in the study will be obtained. Patients will then be followed and managed according to routine care (visits and examinations).

Routine care includes:

* A clinical assessment of efficacy and safety at weeks 12, 24, 36, 52, and 104;
* Oral prednisone treatment at the initial doses recommended by international and French guidelines, in accordance with routine care.

Treatment with upadacitinib will be initiated at the time of patient inclusion (one 15 mg tablet per day) and will be maintained for 104 weeks. Data will then be collected from the participant's medical record (including medical reports, original laboratory test results, imaging reports and medical examinations, and nursing records) for the period of participation in the research, solely for the purpose of meeting the objectives of the research. Clinical, biological, and radiological efficacy data, as well as treatment safety, will be prospectively analyzed at 3, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

Patients aged over 18 years; Signed informed consent; Affiliation with the French national social security system; Diagnosis of newly diagnosed or relapsing GCA according to the 2022 ACR/EULAR criteria; Active aortitis related to GCA demonstrated by imaging (CT angiography, MR angiography, and/or PET-CT); Indication for treatment with an anti-JAK agent within the scope of the marketing authorization for GCA: failure of, intolerance to, or contraindication to tocilizumab therapy; No contraindication to JAK inhibitors.

Exclusion Criteria:

* Pregnancy or breastfeeding (for women of childbearing potential, a negative serum pregnancy test will be required); History of severe immunosuppression, HIV infection, hepatitis C virus (HCV), or positive hepatitis B surface antigen (HBsAg); Non-response to or intolerance of a previous anti-JAK treatment; Positive QuantiFERON test (QFT-TB Gold In-Tube) indicating active tuberculosis (latent tuberculosis under treatment for at least 3 weeks may be included); Receipt of live vaccines within the 3 months preceding treatment initiation; History of malignancy within the past 5 years; Severe renal impairment (creatinine clearance < 30 mL/min/1.73 m²); Hepatic dysfunction defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≥ 5 times the upper limit of normal;

Abnormal blood counts:

Platelets < 50 × 10³/mm³; Neutropenia < 1,000/mm³; Hemoglobin < 8 g/dL; History of thromboembolic disease; History of severe cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with giant cell arteritis (GCA) and active aortitis, with an indication for treatment with an anti-JAK agent within the scope of the marketing authorization for GCA.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving remission of GCA | Week 24.
  the proportion of patients achieving remission of GCA at week 24.

SECONDARY OUTCOMES:
Cumulative incidence of relapses | Weeks 12, 24, 36, 52, and 104;
  Cumulative incidence of relapses at weeks 12, 24, 36, 52, and 104;
Cumulative incidence of GCA remission according to the EULAR consensus definitions | Weeks 12, 36, 52, and 104;
  Cumulative incidence of GCA remission according to the EULAR consensus definitions at weeks 12, 36, 52, and 104;
Cumulative prednisone dose | Weeks 12, 24, 36, 52, and 104;
  Cumulative prednisone dose at weeks 12, 24, 36, 52, and 104;
Cumulative incidence of adverse events and serious adverse events | Weeks 12, 24, 36, 52, and 104
  Cumulative incidence of adverse events and serious adverse events at weeks 12, 24, 36, 52, and 104
Proportion of aortic inflammatory activity as well as radiological vascular progression (i.e., new aortic dilatation and/or stenosis) | Weeks 24, 52, and 104,
  Proportion of aortic inflammatory activity as well as radiological vascular progression (i.e., new aortic dilatation and/or stenosis) at weeks 24, 52, and 104, assessed by CT angiography, MR angiography, and/or PET-scan;
Cumulative incidence rate of the need for vascular, endovascular, or surgical revascularization procedures due to inflammatory activity | Weeks 24, 52, and 104.
  Cumulative incidence rate of the need for vascular, endovascular, or surgical revascularization procedures due to inflammatory activity at weeks 24, 52, and 104.

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Clinique Axium - Aix-en-provence, Aix-en-Provence
  - CHU Caen Normandie, Caen
  - CHU de Dijon, Dijon
  - CH du Mans, Le Mans
  - APHM_Hôpital Nord, Marseille
  - APHM_Hôpital La Conception, Marseille
  - GHSIF Melun, Melun
  - GHI Le Raincy Montfermeil, Montfermeil
  - CHU Nantes - Hotel-Dieu, Nantes
  - APHP_Hôpital St Antoine, Paris
  - APHP_ Hôpital Pitié-Salpêtrière, Paris
  - CHU Rouen_Hôpital Charles Nicolle, Rouen
  - APHP_Hopital Lariboisière, Paris, Île-de-France Region
  - APHP_Hôpital Bichat, Paris, Île-de-France Region